CLINICAL TRIAL: NCT02804646
Title: Recombinant Human Endostatin Durative Transfusion Combined With Pemetrexed Plus Cisplatin or Carboplatin in the First-line Treatment of Advanced Lung Adenocarcinoma With Wild-type EGFR or ALK-negative
Brief Title: Endostar Durative Transfusion Combined With Chemotherapy in the Treatment of Advanced Lung Adenocarcinoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20160606
Record Dates: First submitted 2016-06-15; First posted 2016-06-17 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Adenocarcinoma of Lung
Keywords: Recombinant human endostatin(Endostar); Durative transfusion; adenocarcinoma of lung
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — Endostatins; endostar protein; Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- endostar and chemotherapy group (Experimental): recombinant human endostatin(endostar) injection was continuous intravenous transfusion for 7 days,with the dose of 15mg/m2 per one day,every 21 days of a cycle,combined with pemetrexed plus cisplatin or carboplatin.
  Interventions: Drug: recombinant human endostatin; Drug: pemetrexed plus cisplatin or carboplatin
- chemotherapy group (Active Comparator): pemetrexed injection was intravenous with the dose of 500mg/m2 on day 1 of every 21 days,plus cisplatin or carboplatin,without recombinant human endostatin.
  Interventions: Drug: pemetrexed plus cisplatin or carboplatin

INTERVENTIONS:
Drug: recombinant human endostatin — endostar was continuous intravenous transfusion for 7 days，with the dose of 15mg/m2 for one day
  Other Names: endostar
  Arms: endostar and chemotherapy group
Drug: pemetrexed plus cisplatin or carboplatin — the dose of pemetrexed was 500mg/m2 on day 1 of every 21 days,plus cisplatin or carboplatin.
  Other Names: pemetrexed disodium

SUMMARY:
The purpose of this study is to discuss the efficacy and safety of recombinant human endostatin(endostar) durative intravenous transfusion combined with pemetrexed plus cisplatin or carboplatin in the first-line treatment of advanced lung adenocarcinoma with wild-type EGFR or ALK-negative,compared with chemotherapy without endostar.

DETAILED DESCRIPTION:
With the progress of molecular biology and translational medical research, the treatment of advanced non-small cell lung cancer goes into the era of personalized medicine. Lung adenocarcinoma accounts for about 50% of non-small cell lung cancer.In recent years, although individualized targeted therapy in lung adenocarcinoma progress by leaps and bounds, but the research of wild-type EGFR or ALK-negative lung adenocarcinoma is extremely lag, lack of clinically effective targeted drugs.As time goes on,almost all of the EGFR-TKI treatment of lung adenocarcinoma will be resistant one day,and patients need other treatments, such as chemotherapy.Currently, chemotherapy is still the main treatment for advanced lung adenocarcinoma with EGFR wild-type and unkown.Many researches has reported that:endostar combined with chemotherapy in patients with advanced NSCLC can significantly improve the patient's RR,TTP and did not increase the adverse effects of chemotherapy.Recently,endostar durative intravenous transfusion has been widely accept and use because of the lower toxicity.The purpose of our study was to discuss the efficacy and safety of endostard durative intravenous transfusion combined with chemotherapy.In our study,Patients with Ⅲb/Ⅳ lung adenocarcinoma were divided into two groups randomly,one group was treated with endostar durative intravenous transfusion combined with chemotherapy,while the other group with chemotherapy pemetrexed plus cisplatin or carboplatin only.In the end,PFS,ORR,DCR and OS were compared between these two groups.

ELIGIBILITY:
Inclusion Criteria:

* 1) histologically confirmed (patients not receiving a single sputum cytology diagnosis) non-small cell lung cancer patients,with wild-type EGFR and ALK-negative; 2) According to IASLC2009 new TNM staging of lung cancer stage ⅢB or Ⅳ, previously untreated or relapsed after 1 year of lung cancer resection; 3) have at least one evaluable lesions,according to version 1.1 of the standard in accordance with a judgment RECIST(longest diameter on a spiral CT at least 10mm,on a regular CT longest diameter at least 20mm); 4) Male or female, aged 18 to 75 years; 5) ECOG PS 0 or 1; 6) expected survival at least 3 months; 7) adequate hematological function: absolute neutrophil count (ANC) at least 2×10^9/L and platelet count at least 100×10^9/L and hemoglobin at least 9 g/dL; 8) adequate liver function: total bilirubin less than upper limit of normal (ULN); AST and ALT less than 2.5 times upper limit of normal (ULN); alkaline phosphatase less than 5 times the upper limit of normal (ULN); 9) adequate renal function: serum creatinine less than upper limit of normal (ULN) or calculated creatinine clearance at least 60 mL/min; 10) ECG is normal, there is no non-healing wounds on the body; 11) had not received previous treatment anticancer drugs, or had only received for previous non-metastatic tumors adjuvant or neoadjuvant chemotherapy, but when you start to study treatment has ended more than 6 months; 12) have conducted previous surgery patients required to study treatment was started more than four weeks, and the patient had recovered; 13) have an intact uterus in women prior to enrollment in the study must have a negative pregnancy test result (unless it is already 24 months of amenorrhea) within 28 days. If the pregnancy test from the first administration more than seven days, urine pregnancy test is required for authentication (less than 7 days before the first dose); 14) previous to biological agents, particularly E.coli genetically engineered products without serious allergic reactions; 15) signed informed consent.

Exclusion Criteria:

* 1) pregnancy, breast-feeding women, or female patients of childbearing potential but did not take contraceptive measures;2) existing severe acute infection and is not controlled; or purulent and chronic infection, delayed healing wounds; 3) the original severe heart disease, including congestive heart failure, uncontrolled high-risk arrhythmias, unstable angina, myocardial infarction, severe heart valve disease and resistant hypertension; 4) suffering from neurological and psychiatric diseases or mental disorders is not easy to control, poor compliance, and can not be described with treatment responders; primary brain or central nervous metastasis disease has not been controlled, with significant cranial hypertension or neuropsychiatric symptoms; 5) have bleeding tendencies; 6) other researchers believe that patients should not participate in the present trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
progression free survival | Throughout the study period，an average of 1.5 year

SECONDARY OUTCOMES:
objective response rate | Throughout the study period，an average of 1.5 year
disease control rate | Throughout the study period，an average of 1.5 year
overall survival | after the study finished，an average of 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Lejie Cao, professor, Principal Investigator — Anhui Provincial Hospital
Locations (1):
- Anhui provincial hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided